CLINICAL TRIAL: NCT07046104
Title: Patient Satisfaction and Oral Health Related Quality of Life for Implant Retained Overdenture VERSUS Implant Canine Retained Overdenture. Crossover Clinical Study.
Brief Title: Implant Retained Overdenture VERSUS Implant Canine Retained Overdenture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A0103024RP
Record Dates: First submitted 2025-01-10; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2023-01

CONDITIONS: Oral Health Impact Profile Short Version 14 (OHIP 14)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- implant retained group (Active Comparator): two implants in molar position and two remaining canines
  Interventions: Other: implant retained overdenture prosthesis
- implant tooth retained group (Active Comparator): implant in molar position and two remaining canines
  Interventions: Other: implant canine retained overdenture prosthesis

INTERVENTIONS:
Other: implant retained overdenture prosthesis — implant retained only prosthesis
  Arms: implant retained group
Other: implant canine retained overdenture prosthesis — prosthesis retention from implant and canine
  Arms: implant tooth retained group

SUMMARY:
ABSTRACT Background: mandibular class 1 modification 1 RPD can be retained by mesially placed implant only, or canines can be used to share in retention using telescopic attachment. So, the aim of this clinical study is to evaluate patient satisfaction and oral health impact profile (OHIP-14) for implant retained Overdenture versus implant-tooth retained Overdenture.

Methods: This clinical cross-over study included 10 partially edentulous patients with only remaining mandibular canines. Every patient received two mandibular implants at the 1st premolar region. Two mandibular implant retained overdenture will be constructed, opposing a maxillary single denture. One of the dentures was made with a design based on implant retention only but the other denture was made with dual implant-tooth retention design. The effects of each overdenture design were evaluated after 3 months. patients indicated satisfaction with their prosthesis using a visual analog scale (VAS)Regarding VAS, participants were asked to score their answer according to the amount of satisfaction on a 100 mm line (Score 0 = no satisfaction at all and score 100 = complete satisfaction). The questions cover several items related to overdentures such as retention, stability, comfort, ease of cleaning, ease of speaking, ease of chewing, limited activities due to embarrassment, quality of bolus, and appearance. , and oral health impact profile (OHIP-14) was recorded for both prostheses. The Wilcoxon signed-rank test was done to compare the statistically significant difference between the two groups. SPSS ver.23. P <.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* This research will be done on patients who were previously received 2 mesially placed implants in the 1st premolar region with only two remaining mandibular canines with opposing maxillary single denture

Exclusion Criteria:

* uncontrolled diabetic patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
patients indicated satisfaction with their prosthesis using a visual analog scale (VAS) | 3 months

SECONDARY OUTCOMES:
oral health impact profile (OHIP-14) was recorded for both prostheses. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Basmsa, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided